CLINICAL TRIAL: NCT05586074
Title: HEC73543 Versus Salvage Chemotherapy in Relapsed or Refractory FLT3-ITD Acute Myeloid Leukemia: a Multicenter, Open-label, Randomized Phase 3 Trial
Brief Title: HEC73543 Versus Salvage Chemotherapy in R/R FLT3-ITD AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEC73543-AML-301
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Acute Myeloid (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Azacitidine; Decitabine; Idarubicin; Ida-FLAG protocol; Granulocyte Colony-Stimulating Factor; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clifutinib (Experimental): Subjects received 40 mg dose orally once a day in continuous 28-day cycles, at least 2 hours before and after food. Clifutinib treatment continued until sujects met one of the treatment discontinuation criteria.
  Interventions: Drug: Clifutinib
- Salvage Chemotherapy (Active Comparator): Subjects received chemotherapy in 28-day cycles. Subjects on Low-Dose Cytarabine (LoDAC) received 10 mg of cytarabine twice daily by subcutaneous (SC) or intravenous (IV) injection for 10~14 days. Subjects on azacitidine received 75 mg/m^2 daily by SC for 7 days. Subjects on decitabine received 20 mg/m^2 daily by IV injection for 5 days. Subjects on LoDAC or azacitidine or decitabine treatment continued until they met discontinuation criteria. Subjects on Ara-C±IDA chemotherapy received cytarabine 1~3 g/m^2 daily by IV for 3 days and idarubicin 10 mg/m^2 daily by IV for 3 days. Participants on FLAG-IDA chemotherapy received G-CSF 300 μg/m^2 daily by SC for 6 days (days 1-6), fludarabine 30 mg/m^2 daily by IV for 5 days (days 2-6), cytarabine 1~2 g/m^2 daily by IV for 5 days (days 2-6) and idarubicin 10 mg/m^2 daily by IV for 3 days (days 2-4). Subjects receiving Ara-C±IDA or FLAG-IDA received 1 cycle of therapy and were assessed for response on day 28+/-2 days.
  Interventions: Drug: LoDAC; Drug: Azacitidine; Drug: Decitabine; Drug: Ara-C±IDA; Drug: FLAG-IDA

INTERVENTIONS:
Drug: Clifutinib — tablet, oral
  Other Names: HEC73543
  Arms: Clifutinib
Drug: LoDAC — subcutaneous (SC) or intravenous (IV) injection
  Other Names: Low Dose Cytarabine
  Arms: Salvage Chemotherapy
Drug: Azacitidine — SC or IV
  Arms: Salvage Chemotherapy
Drug: Decitabine — IV
  Arms: Salvage Chemotherapy
Drug: Ara-C±IDA — SC and IV
  Other Names: Cytarabine, Idarubicin
  Arms: Salvage Chemotherapy
Drug: FLAG-IDA — SC and IV
  Other Names: Granulocyte-Colony Stimulating Factor (G-CSF), Fludarabine, Cytarabine, Idarubicin
  Arms: Salvage Chemotherapy

SUMMARY:
A randomized，multicenter, open-label Phase III, clinical study is conducted to evaluate the clinical benefit Clifutinib in Chinese patients with relapsed/ refractory (R/R) FLT3-mutated AML as shown with overall survival compared to salvage chemotherapy, and also to investigate the efficacy of Clifutinib as assessed by CR/CRh rate in these subjects.

DETAILED DESCRIPTION:
Subjects who are at least 18 years and above at the time of signing informed consent may participate in this study. Subjects will be randomized in a 2:1 ratio to receive Clifutinib or salvage chemotherapy. Subjects will enter the screening period up to 28 days prior to the start of treatment. Prior to randomization, a salvage chemotherapy regimen will be pre-selected for each subjects; options will include low-dose cytarabine (LoDAC), azacitidine, decitabine, Ara-C±IDA or FLAG±IDA. The randomization will be stratified by response to first-line therapy and pre-selected salvage chemotherapy. Participants will be administered treatment over continuous 28-day cycles.

After treatment discontinuation, participants will have a end-of-treatment visit within 7 days after treatment discontinuation, followed by a 30-day follow-up for safety. After that, long term follow-up will be done every 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at the time of obtaining informed consent.
* Subject has a diagnosis of primary acute myeloid leukemia (AML) or AML secondary to myelodysplastic syndrome (MDS) according to WHO classification;
* Subject is refractory to or relapsed after first-line AML therapy (with or without hematopoietic stem cell transplant )
* Subject is positive for FLT3 mutation in bone marrow or whole blood as determined by the central lab
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subject is eligible for pre-selected salvage chemotherapy at the investigator's discretion

Exclusion Criteria:

* Subject has received prior treatment with other FLT3 inhibitors
* Subject has AML that has relapsed after or is refractory to more than 1 line of therapy
* Subject has an active uncontrolled infection
* Subject is known to have human immunodeficiency virus infection
* Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
OS | From the date of randomization until the date of death from any cause, assessed up to 5 years
  Overall survival was defined as the time from the date of randomization until the date of death from any cause
CR/CRh rate | From randomization until the data cut-off date of April 2025, all subjects included in the primary analysis of CR/CRh rate were followed up at least 4 months
  The CR/CRh rate was defined as the number of subjects who achieved either CR or CRh at any of the postbaseline visits divided by the number of subjects in the analysis population

SECONDARY OUTCOMES:
EFS | From randomization until the data cut-off date of June 2026, median time of follow-up for OS was 15 months
  EFS was defined as the time from the date of randomization until the date of documented relapse, treatment failure, new anti-leukemia therapy or death from any cause
CR rate | From randomization until the data cut-off date of June 2026, all subjects included in the analysis of CR rate were followed up at least 4 months
  The CR rate was defined as the number of subjects who achieved the best response of CR divided by the number of subjects in the analysis population
CRc Rate | From randomization until the data cut-off date of June 2026, all subjects included in the analysis of CRc rate were followed up at least 4 months
  CRc rate was defined as the number of subjects who achieved the best response of CRc (CR, CRh or CRi divided by the number of subjects in the analysis population
Adverse Events | From ICF signature date up to 30 days after the last dose of study drug, median treatment duration for Clifutinib was 140 days versus salvage chemotherapy 140 days
  Number of Participants With Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- the First Affiliated Hospital,College of Medicine,Zhejiang University, Hanzhou, China

IPD SHARING:
Plan to Share IPD: No